CLINICAL TRIAL: NCT06604975
Title: Arginin-stimulated Copeptin in Polyuria-polydipsia Syndrome in Children
Acronym: COPEPCHILD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM23_0379
Record Dates: First submitted 2024-09-09; First posted 2024-09-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Primary Polydipsia; Central Diabetes Insipidus; Nephrogenic Diabetes Insipidus
MeSH Terms: conditions — Polydipsia, Psychogenic; Diabetes Insipidus, Neurogenic; Diabetes Insipidus, Nephrogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NDI-PP- CDI groups (Experimental): Copeptin represents a new biomarker, direct mirror of AVP release with remarkable characteristics (stable, rapid determination, small blood volume). Copeptin has become a diagnostic tool in adult PPS and eliminated WDT in the diagnostic process. In children, basal copeptin values help for NDI and to exclude CDI (basal copeptin threshold > 30 and >3.53 pmol/l (Se 100%, Sp 87.4%), respectively). Below 3.53 pmol/l, basal copeptin performance was inadequate to discriminate PP and CDI, highlighting the relevance of the stimulated copeptin study to improve this strategy.
  Interventions: Procedure: Measure of Basal Copeptin level; Procedure: Measure of arginine-stimulated copeptin; Procedure: IRM; Behavioral: Water reduction at home

INTERVENTIONS:
Procedure: Measure of Basal Copeptin level — Copeptin test is performed after solid fasting since midnight without water restriction. After blood collection on heparin tube used for biological inclusion criteria, heparinized plasma is transferred to Timone University hospital (transport temperature +4°C) for screening copeptin assay.
  The basal copeptin level determines the next step:
  1. copeptin ≥ 30 pmol/L defines the diagnosis of NDI and results in a specific care;
  2. copeptin < 30 pmol/L defines the group of eligible patients for arginine stimulation
Procedure: Measure of arginine-stimulated copeptin — The arginine-stimulated copeptin test start at 8 am, after solid fasting since midnight without water restriction, and 30 min of rest in decubitus position. A dose of 0.5 g/kg of arginine (maximum 40g) diluted in 0.9% NaCl is infused over 30 min through a peripheral venous line. Copeptin is measured at T0 (before infusion), T45, T60, T90, and T120 min after infusion.
Procedure: IRM — Based on our previous study, patients with basal copeptin value over 3.53 pmol/L are considered as positive diagnosis of PP (Se 100%, Sp 87.4%) and cerebral MRI is not performed for this group of patients (PP group).
  A cerebral and pituitary MRI performed according to reference procedures (without and with contrast medium used in routine care) for patients considered as an uncertain diagnosis (UD) based on basal copeptin value (< 3.53 pmol/L). MRI interpretation is performed by two independent neuroradiologists (one from the recruiting center and one from the pilot center). In case of discrepancies, a third independent interpretation will be performed by a neuroradiologist from the coordinating center. Abnormal pituitary MRI (thickened pituitary stalk pituitary tumor, ectopic neurohypophysis, septo-optic dysplasia, empty sellar, Rathke pouch) allows a diagnosis of CDI leading to etiological investigations and AVP treatment.
Behavioral: Water reduction at home — Patients with basal copeptin ≥ 3.53 pmol/l (PP group), and UD patients with normal MRI have gradual reduction of water intake at home without AVP treatment : gradual reduction with 20% in the first week, 30% in the second, 40% in the third, reaching 50% of daily fluid in the last week including restriction overnight, deletion drink before sleep. Some recommendations will be provided to help physicians. For all these latest patients, a clinical reassessment (weight, height, heart rate, blood pressure, input/output 24 hours balance) is performed one month later.

SUMMARY:
The exploration of polyuro-polydipsia syndrome (PPS) with hypotonic polyuria should distinguished, primary polydipsia (PP) due to excessive water intake, central diabetes insipidus (CDI) related to insufficient secretion of antidiuretic hormone (AVP), and nephrogenic diabetes insipidus (NDI) related to AVP insensitivity. The determination of plasma AVP is not relevant (unstable concentration, short in vitro half-life, long technical time and large blood sample). The differential diagnosis is currently based on a water deprivation test (WDT), an indirect reflection of AVP action, requiring more than 6 hours of hospitalization with risk of dehydration and low accuracy. Copeptin represents a new biomarker, direct mirror of AVP release with remarkable characteristics (stable, rapid determination, small blood volume). Copeptin has become a diagnostic tool in adult PPS and eliminated WDT in the diagnostic process. In children, basal copeptin values help for NDI and to exclude CDI (basal copeptin threshold > 30 and > 3.53 pmol/l (Se 100%, Sp 87.4%), respectively). Below 3.53 pmol/l, basal copeptin performance was inadequate to discriminate PP and CDI, highlighting the relevance of the stimulated copeptin study to improve this strategy. The arginine stimulation test is widely used as a simple, short duration (2 hours) and well tolerated tool to diagnose growth hormone deficiency in pediatrics. The performance of this test for copeptin stimulation was studied in adults with PPS with a high diagnostic accuracy.

The aim of the study is identify the best discriminant threshold of the arginine stimulation test in the uncertain diagnosis (basal copeptin <30 pmol/l) in the polyuro-polydipsic syndrome in children.

Then evaluate the discriminative capacities of the arginine stimulation test between the primary polydipsia and central insipid diabetes in the polyuro-polydipsic syndrome in children. And finally evaluate the cost-effectiveness of a new decisional algorithm for the differential diagnosis of PPS in children and evaluate the impact of infusion volume on copeptin secretion using the protidemia copeptin ratio.

DETAILED DESCRIPTION:
Routine biochemical tests are performed to screen patients for PPS and determine basal copeptin level after solid fasting since midnight without water restriction: 1/ a basal copeptin value ≥ 30 pmol/L defines the diagnosis of NDI and results in a specific care; 2/ a basal copeptin < 30 pmol/L defines the group of eligible patients for arginine stimulation. The arginine-stimulated copeptin test start at 8 am, at the dose of 0.5 g/kg over 30min. Copeptin is measured at T0 (before infusion), T45, T60, T90, and T120 min after infusion.

Patients with basal copeptin value over 3.53 pmol/L are considered as positive diagnosis of PP (Se 100%, Sp 87.4%) and cerebral MRI is not performed for this group of patients (PP group).

Patients with basal copeptin value < 3.53 pmol/L are considered as an uncertain diagnosis (UD) and cerebral and pituitary MRI is performed with a least two independent interpretations. Abnormal pituitary MRI allows a diagnosis of CDI leading to etiological investigations and AVP treatment. Patients with basal copeptin ≥ 3.53 pmol/l (PP group), and UD patients with normal MRI have gradual reduction of water intake without AVP treatment. For all these latest patients, a clinical and biological reevaluation is performed one month later.

The gold standard will be the final diagnosis PP vs. CDI based on a set of indicators: medical history, physical examination, pituitary hormonal assessment, hypothalamo-pituitary MRI, follow-up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 18 years with polyuro-polydipsia syndrome (defined as hypotonic diuresis > 50 mL/kg/day in pediatric age or 30 mL/kg/day in late puberty (Tanner 5)) presenting for differential diagnosis between PP and DIC
* Basal copeptin of less than 30 pmol/l
* Agreeing to participate in the study
* Whose two parents' consent to have their child participate in the study.

Exclusion Criteria:

* Diabetes mellitus
* Unbalanced dysthyroidism
* Corticotropic deficiency
* Ionic disorders (dysnatremia < 135 or > 145 mmol/l, dyskalemia < 3 or > 5 mmol/l, corrected dyscalcemia < 2.2 or > 2.6 mmol/L)
* Moderate to severe clinical dehydration (recent weight loss > 5% of body weight, clinical or biological signs of dehydration) requiring immediate therapeutic management
* Renal failure with GFR < 60 mL/min/1.73 m2
* Uropathy
* Tumor syndrome (except hypothalamo-pituitary tumor)
* Intracranial hypertension
* ROHHAD syndrome
* Fever or biological inflammatory syndrome with CRP > 5 mg/L
* Hepatic insufficiency
* Contraindication to MRI
* Contraindication to progressive water intake restrictions
* History of contraindication to arginine
* Positive test for Pregnancy
* Lack of authorization by both parents or legal representatives

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of arginine-stimulated copeptine level | Different time points of argenine stimulates copeptine level will be measured at 45 minutes, 60 minutes, 90 minutes and 120 minutes
  Determine arginine-stimulated copeptine level for each time (T45min, T60min, T90min, T120min)

SECONDARY OUTCOMES:
Cost savings applying a new algorithm for the exploration of the Polyuria-polydipsia Syndrome using an Argenin-stimulated copeptin test | Month 36
  Evaluate the cost-effectiveness of a new decisional algorithm for the differential diagnosis of PPS in children including medications, examinations and length of stay at the hospital
Copeptin Ratio | Month 36
  Evaluate the impact of infusion volume on copeptin secretion using the copeptin ratio (for each time, the arginine-stimulated copeptin ratio will be calculated in order to take count of the baseline copeptin concentration and in order to counteract any blood dilution due to perfusion copeptin ratio will be corrected by protidemia)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel REYNAUD, Pr, Principal Investigator — AP-HM
Locations (14):
- France (14):
  - CHU Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU Lille, Lille
  - HCL, Lyon
  - Assistance Publique Hopitaux de Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - AP-HP, Paris
  - CH Pau, Pau
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No